CLINICAL TRIAL: NCT03503708
Title: Antioxidant for Improvement of Hepatic Function in Patients With Alcohol Liver Disease Without Cirrhosis: Non-randomized Interventional Cohort Study
Brief Title: Herbal Supplements for Improvement of Liver Function in Participants With Alcoholic Liver Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Composite Interceptive Med Science (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OI-009-2018
Record Dates: First submitted 2018-04-11; First posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Alcoholic Liver Disease
MeSH Terms: conditions — Liver Diseases, Alcoholic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): All the eligible participants will receive Livitol-17 capsules. It consist of 390 mg of whole herbs and extract of Phyllanthus niruri (Bhumyamalaki), Boerhaavia diffusa (Punarnava) and Picroorrhiza kurroa (Katuki).
  Interventions: Drug: Livitol-70

INTERVENTIONS:
Drug: Livitol-70 — Livitol-17 detoxifies, purifies and rejuvenates liver, kidney and spleen. Participants will be given the intervention in two bottles at each visit. Participant will be instructed to take two capsule twice daily at a fixed time in the day.

SUMMARY:
Alcoholic liver disease represents the major health issues and it ranges from simple steatosis to cirrhosis. There is a paucity of data to support the allopathic intervention among these group of patients. Livitol-17 consist of the 3 whole herbs and extract which has antioxidant, hepatoprotective as well as reno-protective properties. The aim of this trial is to study the efficacy of herbal supplement to improve the liver function of alcoholic liver disease subject.

ELIGIBILITY:
Inclusion Criteria:

Adults aged over 18 years with the evidence of alcoholic liver disease (ALD) based on a thorough history, physical examination, and laboratory tests and all of the following:

* Chronic alcohol intake, Identified with AUDIT(Alcohol Use Disorder Inventory Test) Questionnaire
* Active alcohol use until 4 weeks prior to presentation
* ALT and AST elevated >1.5 times the upper limit of normal
* Over 1.5 ratio of AST to ALT
* Maddrey Discriminant function(DF) less than 30

Exclusion Criteria:

* Severe alcoholic hepatitis with cirrhosis or life expectancy less than 3 months
* Severe renal impairment (Glomerular filtration rate below 60 ml/min per 1.73m2)
* Hepatic disorders due to cardiac causes, inherited metabolic causes, hemochromatosis and Wilson's disease
* Participants with active viral hepatitis
* Under going active treatment for alcohol withdrawal syndrome(AWS) at the study entry
* Participants on hepatotoxic medications like antitubercular medication, antiviral medication, paracetamol etc.
* Pregnant, attempting to conceive, or lactating women
* Participating in another clinical trial with an active intervention or drug or device with last dose taken within 60 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-05-30 (Estimated); Primary Completion 2018-10-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in AST(Aspartate Aminotransferase) | 3 months
  The above mentioned test will be measured with panel of Liver function test at central laboratory.
Change from baseline in ALT(Alanine Aminotransferase) | 3 months
  The above mentioned test will be measured with panel of Liver function test at central laboratory.
Change from baseline in ALP(Alkaline Phosphatase) | 3 months
  The above mentioned test will be measured with panel of Liver function test at central laboratory.
Change from baseline in GGT(Gamma Glutamyl Transferase) | 3 months
  The above mentioned test will be measured with panel of Liver function test at central laboratory.
Change from baseline in serum total bilirubin | 3 months
  The above mentioned test will be measured with panel of Liver function test at central laboratory.
Number of Subject with adverse events | 3 months
  Adverse events is defined as any untoward medical occurrence that may not necessarily have a causal relationship with the treatment, but resulted in a dose reduction or discontinuation of treatment.

SECONDARY OUTCOMES:
Change in radiological response | 3 months
  The degree of fatty infiltration will be assessed by ultrasound.
Change in maddrey discriminant function(DF) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Alben Sigamani, MD, Principal Investigator — Narayana Hrudayalaya Hospital; Sanjaya Chauhan, PharmD, Study Chair — Composite Interceptive Med Science
Locations (1):
- Mazumdar Shaw Medical Centre, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: Undecided